CLINICAL TRIAL: NCT04446325
Title: Venous Disease Thromboembolic and Amyotrophic Lateral Sclerosis
Acronym: TESLA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0236
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Lateral Amyotrophic Sclerosis; Venous Thrombo-embolic Desease
Keywords: lateral amyotrophic sclerosis; venous thrombo-embolic desase; pulmonary embolism; deep venous thrombosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thrombo-embolic (VTE) rates could be high in patients with amyotrophic lateral sclerosis (ALS). Indeed, the rate of VTE in this specific population could be 7-fold higher in this population. Predictiv factors of VTE in patients with ALS are mobility reduction and neurological paralysis. However, to our knowledge, medical littérature is poor concerning VTE and ALS association.

Our first aim is to define annual rate of VTE in ALS population.Then we aim to identify predictiv factors of VTE in this specific population. The studied population is Brest universitary hospital cohort of ALS patient included between 2000 and 2019.

ELIGIBILITY:
Inclusion Criteria:

* patients with amyotrophic lateral sclerosis defined by revised El Escorial score criteria followed in competence centre of Brest Universitary Hospital during 2000 to 2019

Exclusion Criteria:

* no consent
* other neuro-degenerativ diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with amyotrophic lateral sclerosis defined by revised El Escorial score criteria followed in competence centre of brest universitary hospital during 2000 to 2019
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of venous thrombo-embolic eventsrate per year in amyotrophic lateral sclerosis patients followed between 2000 and 2019 in Brest universitary hospital | 19 years
  pulmonary embolism and deep venous thrombosis

SECONDARY OUTCOMES:
Number of predictiv factors of venous thrombo-embolism events in amyotrophic lateral sclerosis population followed in Brest universitary hospital between 2000 and 2019 | 19 years
  immobilization, impairment of respiratory function,, mecanical ventilation, denutrition, artificial nutrition

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France